CLINICAL TRIAL: NCT01690715
Title: Prognostic Value Related to the Presence of Thrombosis or Portal Vein Invasion in Patients With Hepatocellular Carcinoma Submitted to Surgery
Acronym: HSL2012-06
Status: Terminated | Type: Observational
Why Stopped: There was recruted subject
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Frederico Perego Costa, Attending physician, Hospital Sirio-Libanes
Other Study IDs: HSL 2012/06
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Thrombosis; Hepatic Portal Vein Tumor Invasion
Keywords: Hepatocellular Carcinoma; Thrombosis; Portal Vein Invasion
MeSH Terms: conditions — Carcinoma, Hepatocellular; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hepatocellular carcinoma underwent surgery

SUMMARY:
A retrospective study based on analysis of medical records of patients with hepatocellular carcinoma treated at the Hospital Sírio-Libanês (Sao Paulo-Brazil) between 2001 and 2011 with diagnosis confirmed by imaging or histological specimen underwent surgical resection with curative intent. The study aims to determine the prognostic value of vascular complications related to cancer and to evaluate the survival rate of these patients, comparing the data with those reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma confirmed by imaging or histological specimen underwent surgical resection, with or without hepatic cirrhosis association;
* presence of venous outflow obstruction, either by direct tumor invasion or thrombosis, on portal vein or one of its main vessels;

Exclusion Criteria:

* Patients undergoing prior systemic treatment;
* Patients presenting incomplete data that do not allow their classification according to the stratification models;
* Patients whose information of progression or death can not be recovered;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with hepatocellular carcinoma confirmed by imaging or histological specimen underwent surgical resection with curative intent with the presence of venous outflow obstruction, either by direct tumor invasion or thrombosis, on portal vein or one of its main vessels.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-30 (Actual)

PRIMARY OUTCOMES:
Prognosis (disease graduation) | 1 to 3 years
  The carcinoma prognosis in the presence of vascular complications related to cancer, characterized by invasion or portal vein thrombosis.

SECONDARY OUTCOMES:
Survival rate in years | 1 to 3 years
  Determination of the survival rate within 1 to 3 years for those submitted to curative hepatectomy.
Relation established between survival and degree of underlying liver dysfunction | 1 to 3 years
  Investigate a possible relationship between survival and degree of underlying liver dysfunction in patients with thrombosis or portal vein invasion in patients undergoing curative hepatectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanês, São Paulo, Brazil